CLINICAL TRIAL: NCT06373601
Title: Selution Sirolimus Coated Balloon (MedAlliance) Versus SeQuent Please Neo Paclitaxel Coated Balloon (Bbraun) for the Treatment of de Novo Coronary Artery Lesions in Medium-small Size Vessels.
Brief Title: SPAGO: Sirolimus Paclitaxel Angiographic Gain Objective
Acronym: SPAGO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Evidence per Attività e Ricerche Cardiovascolari ONLUS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPAGO
Record Dates: First submitted 2024-04-04; First posted 2024-04-18 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Coronary Artery Disease; Stenosis Coronary; Coronary Artery Lesion; Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis

STUDY DESIGN:
Intervention Model Description: 140 subjects will be enrolled in a competitive way and 1:1 randomized to receive treatment with either the study device (SelutionTM) or the control device (SeQuent Please NeoTM). Randomization will be stratified according to DCB length: at least 100 patients treated with DCB ≥ 30 mm will be assigned to either SelutionTM or SeQuent Please NeoTM, while a maximum of 40 patients treated with DCB < 30 mm will be assigned to either SelutionTM or SeQuent Please NeoTM. A minimum of 100 subjects treated with DCB ≥ 30 mm is considered necessary to provide an initial evaluation of intramyocardial resistance measurements, due to the lack of literature data on these parameters.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sirolimus-eluting balloon (Selution) (Experimental): DCB angioplasty with a sirolimus-eluting balloon
  Interventions: Device: sirolimus-eluting balloon (Selution)
- paclitaxel-eluting balloon (SeQuent Please Neo) (Active Comparator): DCB angioplasty with a paclitaxel-eluting balloon
  Interventions: Device: paclitaxel-eluting balloon (SeQuent Please Neo)

INTERVENTIONS:
Device: sirolimus-eluting balloon (Selution) — PCI treatment with DCB, in particular sirolimus coated balloon
  Arms: sirolimus-eluting balloon (Selution)
Device: paclitaxel-eluting balloon (SeQuent Please Neo) — PCI treatment with DCB, in particular paclitaxel coated balloon
  Arms: paclitaxel-eluting balloon (SeQuent Please Neo)

SUMMARY:
The objective of the study is to compare angiographic outcomes of Selution sirolimus coated balloon (MedAlliance) versus SeQuent Please Neo paclitaxel coated balloon (Bbraun) for the treatment of de novo coronary artery lesions in medium size vessels (>2.00 mm and ≤3.00 mm) with respect to Net Gain (mm) and Fractional Flow Reserve (FFR) at 12 months follow-up.

DETAILED DESCRIPTION:
This is a prospective, randomized, multicenter, no-profit and post-market study in subjects with small vessels, i.e. at least one de novo lesion in a small vessel (>2.00 mm and ≤3.00). Vessel size is evaluated by visual estimation. It is possible to include only one study lesion per patient. For the purposes of this study, in cases of diffuse coronary artery disease where overlapped DCB are utilized for the treatment of the lesion, this will be considered as a single lesion. In case of a successful predilatation (i.e. no major (type D, E, F) angiographic dissections, residual stenosis ≤ 30% and TIMI flow = 3), the subject will be randomized in a 1:1 fashion to SelutionTM or SeQuent Please NeoTM. Randomization will be stratified according to DCB length (< 30 mm or ≥ 30 mm) in order to include at least 100 patients treated with DCB of 30 mm or longer. Measurements of intramyocardial resistances, after lesion preparation prior to DCB treatment and after DCB treatment (2 measurements), will be limited to a maximum of 100 lesions treated with DCB ≥ 30 mm. Given the lack of literature data on intramyocardial resistance measurements, a minimum of 100 subjects is considered necessary to provide an initial evaluation of these parameters. With a total sample size of 140 patients for the study, it will be allowed to enroll up to 40 patients treated with DCB < 30 mm. Once this limit is reached, only patients treated with DCB ≥ 30 mm will be enrolled while maintaining a 1:1 randomization ratio. During the index procedure, it is possible to treat other not study lesions (if applicable) with any other commercial device (e.g. drug-eluting stent) if they are located in a different epicardial territory than the study target lesion. All not studylesions should be treated prior to study target lesion procedure, and should be successful and uncomplicated.

Follow-up by phone call will occur at 1 and 6 months post-PCI. At 12 months all subjects will perform an angiographic follow up at the same site where the index procedure was performed. Quantitative Coronary Angiography (QCA) assessment will be performed at baseline (pre- and post-procedure) and on follow up angiography by the imaging core lab. FFR assessment will be performed at the time of follow-up angiography.

All subjects must receive dual anti-platelet therapy (DAPT), being aspirin (ASA) and P2Y12 inhibition therapy for at least 1 month after drug coated balloon PCI or according to standard local practice (with the choice of agent left to the discretion of the investigator), followed by ASA monotherapy indefinitely. However, in case the subject had recent ACS or is receiving additional drug-eluting stents, DAPT must be given according to local standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≥18 years
2. Subject with chronic stable angina or stabilized acute coronary syndromes with normal cardiac biomarker values.
3. The subject has at least one de-novo lesion in a small vessel (>2.00 mm and ≤3.00 mm prior to pre-dilatation) with a diameter stenosis between 50% and 99% (prior to pre-dilatation). It is possible to enroll subjects that have a stent previously implanted in the same epicardial territory (main vessel and ramifications) of the target lesion
4. Patients with target lesion to be treated with DCB < 30 mm in length (up to 40 patients) or with DCB ≥ 30 mm in length (at least 100 patients)
5. Able to understand and provide informed consent and comply with all study procedures including 12 months angiographic follow-up
6. Subject must have completed the follow-up phase of any previous study

Exclusion Criteria:

1. Subject is a woman who is pregnant or nursing (a pregnancy test must be performed within 7 days prior to the index procedure in women of child-bearing potential)
2. Evidence of ongoing acute myocardial infarction (AMI) in ECG and/or elevated cardiac biomarkers (according to local standard hospital practice) have not returned within normal limits at the time of procedure
3. Known contraindication or hypersensitivity to sirolimus, paclitaxel, or to medications such as aspirin, heparin, and all of the following four medications: clopidogrel bisulfate, ticlopidine, prasugrel, ticagrelor
4. Subjects who experienced a previous PCI with DCB in the epicardial territory (main vessel and ramifications) where the target lesion is located, during the last 12 months
5. Subject suffered from stroke/TIA during the last 6 months
6. LVEF <30%
7. Platelet count <100,000 cells/mm3 or >400,000 cells/mm3, a WBC of <3,000 cells/mm3, or documented or suspected liver disease (including laboratory evidence of hepatitis)
8. Known renal insufficiency (e.g. serum creatinine >2,5 mg/dL, creatinine clearance ≤30 mL/min or eGFR ≤30 mL/min/m2), or subject on dialysis, or acute kidney failure (as per physician judgment)
9. Subject undergoing planned surgery within 1 month with the necessity to stop DAPT
10. History of bleeding diathesis or coagulopathy
11. The subject is a recipient of a heart transplant
12. Concurrent medical condition with a life expectancy of less than 12 months
13. The subject is unwilling/not able to return for angiographic re-catheterisation at 12 months follow-up
14. Currently participating in another trial

    Angiographic exclusion criteria:
15. Target vessel size >3.00 mm
16. Target vessel size ≤2.00 mm
17. Target lesion has a diameter stenosis < 50% prior to pre-dilatation
18. Target lesion has a total occlusion or TIMI flow < 2 prior to pre-dilatation
19. Pre-dilatation of the target lesion not performed or not successful (residual stenosis > 30%, TIMI flow < 3 and presence of major angiographic dissections)
20. Target lesion in left main stem
21. The target vessel contains visible thrombus
22. Aorto-ostial target lesion (within 3 mm of the aorta junction)
23. Lesion is located within an arterial or saphenous vein graft or distal to a diseased arterial or saphenous vein graft

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-09-05 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
In-segment (balloon treated area) Net Gain (mm) at 12 months post-procedure | 12 months post-procedure
  The primary endpoint is in-segment (balloon treated area) Net Gain (mm) at 12 months post-procedure. Net Gain is defined as acute gain at the time of the index procedure minus late loss at the time of follow-up angiography.
Fractional Flow Reserve (FFR) | From enrollment to the end of treatment at 12 months
  FFR (absolute value) at 12 months post-procedure

SECONDARY OUTCOMES:
Device success (lesion based) | 12 months post-procedure
  Successful delivery and inflation within 45 seconds of the allocated DCB device at the intended target lesion during an attempt with a DCB not previously used (first use) and successful withdrawal of the device system with attainment of final in-lesion residual stenosis of <30%. I
Procedure success | 12 months post-procedure
  Successful delivery and inflation within 45 seconds of the allocated DCB device at the intended target lesion during an attempt with a DCB not previously used (first use) and successful withdrawal of the device system with attainment of final in-lesion residual stenosis of <30 % without the occurrence of TLF during the index procedure hospital stay).
Angiographic outcomes 1 | 12 months post-procedure
  late lumen loss
Angiographic outcomes 2 | 12 months post-procedure
  minimal lumen diameter
Angiographic outcomes 3 | 12 months post-procedure
  percent diameter stenosis
Angiographic outcomes 4 | 12 months post-procedure
  restenosis rate
Device oriented Composite Endpoint (DoCE/ TLF) | 12 months post-procedure
  DoCE/ TLF which is composite of cardiac death, TV-MI, and clinically indicated target lesion revascularization (TLR)
Acute/subacute/early/late vessel thrombosis | 12 months post-procedure
  Thrombosis should be reported as a cumulative value at the different time points and with the different separate time points. Time 0 is defined as the time point after the guiding catheter has been removed and the patient left the catheterization lab.
Periprocedural myocardial infarction | From enrollment to the end of treatment at 12 months
  Periprocedural myocardial infarction according to the Fourth Universal definition of Myocardial Infarction
PCI related myocardial injury | From enrollment to the end of treatment at 12 months
  PCI related myocardial injury, defined according to the Fourth Universal definition of Myocardial Infarction estimating the absolute value of troponin pre-discharge or within 3-8 hours post-PCI
Absolute difference in CFR for the first 100 patients treated with DCB ≥ 30 mm | baseline
  Absolute difference in CFR measured with a dedicated system (PressureWire™ X Guidewire and Coroventis CoroFlow Cardiovascular System, Abbott)
Absolute variation in IMR for the first 100 patients treated with DCB ≥ 30 mm | baseline
  Absolute variation in IMR from the first assessment (after predilation) to the second assessment (after DCB angioplasty)
Absolute decrease in CFR for the first 100 patients treated with DCB ≥ 30 mm | baseline
  Absolute decrease in CFR from the first assessment (after predilatation) to the second assessment (after DCB angioplasty)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio AC Colombo, MD, Study Chair — Fondazione Evidence ONLUS
Locations (10):
- Italy (10):
  - Clinica Montevergine, Mercogliano, Italy/Avellino
  - ASST Papa Giovanni XXIII, Bergamo, Italy/Bergamo
  - Fondazione Poliambulanza, Brescia, Italy/Brescia
  - Azienda Ospedaliero Universitaria di Ferrara, Ferrara, Italy/Ferrara
  - Centro Cardiologico Monzino, Milan, Italy/Milano
  - Istituto Clinico Humanitas, Rozzano, Italy/Milano
  - Clinica Mediterranea, Napoli, Italy/Napoli
  - Azienda Ospedaliero Universitaria San Luigi Gonzaga, Orbassano, Italy/Torino
  - Ospedale di Rivoli, Rivoli, Italy/Torino
  - Ospedale Sant'Andrea, Vercelli, Italy/Vercelli

REFERENCES:
- [Background] Duan Y, Wang Y, Zhang M, Li Z, Chen L, Miao H, Pei S, Lu Y, Wang Z. Computational Pressure-Fluid Dynamics Applied to Index of Microcirculatory Resistance, Predicting the Prognosis of Drug-Coated Balloons Compared With Drug-Eluting Stents in STEMI Patients. Front Physiol. 2022 May 24;13:898659. doi: 10.3389/fphys.2022.898659. eCollection 2022. PMID 35685283
- [Background] Nishi T, Murai T, Ciccarelli G, Shah SV, Kobayashi Y, Derimay F, Waseda K, Moonen A, Hoshino M, Hirohata A, Yong ASC, Ng MKC, Amano T, Barbato E, Kakuta T, Fearon WF. Prognostic Value of Coronary Microvascular Function Measured Immediately After Percutaneous Coronary Intervention in Stable Coronary Artery Disease: An International Multicenter Study. Circ Cardiovasc Interv. 2019 Sep;12(9):e007889. doi: 10.1161/CIRCINTERVENTIONS.119.007889. Epub 2019 Sep 6. PMID 31525096
- [Background] Fearon WF, Balsam LB, Farouque HM, Caffarelli AD, Robbins RC, Fitzgerald PJ, Yock PG, Yeung AC. Novel index for invasively assessing the coronary microcirculation. Circulation. 2003 Jul 1;107(25):3129-32. doi: 10.1161/01.CIR.0000080700.98607.D1. Epub 2003 Jun 23. PMID 12821539
- [Background] Del Buono MG, Montone RA, Camilli M, Carbone S, Narula J, Lavie CJ, Niccoli G, Crea F. Coronary Microvascular Dysfunction Across the Spectrum of Cardiovascular Diseases: JACC State-of-the-Art Review. J Am Coll Cardiol. 2021 Sep 28;78(13):1352-1371. doi: 10.1016/j.jacc.2021.07.042. PMID 34556322
- [Background] Colleran R, Harada Y, Kufner S, Giacoppo D, Joner M, Cassese S, Ibrahim T, Laugwitz KL, Kastrati A, Byrne RA. Changes in high-sensitivity troponin after drug-coated balloon angioplasty for drug-eluting stent restenosis. EuroIntervention. 2017 Oct 20;13(8):962-969. doi: 10.4244/EIJ-D-16-00939. PMID 28134126
- [Background] Ikenaga H, Kurisu S, Ishibashi K, Dohi Y, Fukuda Y, Kihara Y. Slow-flow phenomenon after Paclitaxel-coated balloon angioplasty: findings from optical coherence tomography and coronary angioscopy. JACC Cardiovasc Interv. 2015 Apr 20;8(4):e59-62. doi: 10.1016/j.jcin.2014.11.016. Epub 2015 Mar 26. No abstract available. PMID 25819189
- [Background] Young M, Cuculi F, Erne P. PTCA with drug-coated balloons is associated with immediate decrease of coronary flow reserve. Catheter Cardiovasc Interv. 2013 Mar;81(4):682-6. doi: 10.1002/ccd.23502. Epub 2013 Jan 29. PMID 23361864
- [Background] Aihara K, Torii S, Ito M, Koseki K, Shiozaki M, Sato Y, Nakamura N, Yoshikawa A, Ikari Y, Nakazawa G. Biological differences of three paclitaxel- and sirolimus-coated balloons on coronary lesions in a rabbit model. EuroIntervention. 2024 Mar 18;20(6):e389-e398. doi: 10.4244/EIJ-D-23-00425. PMID 38506736
- [Background] Kawai K, Rahman MT, Nowicki R, Kolodgie FD, Sakamoto A, Kawakami R, Konishi T, Virmani R, Labhasetwar V, Finn AV. Efficacy and Safety of Dual Paclitaxel and Sirolimus Nanoparticle-Coated Balloon. JACC Basic Transl Sci. 2024 May 1;9(6):774-789. doi: 10.1016/j.jacbts.2024.02.002. eCollection 2024 Jun. PMID 39070273
- [Background] Boitet A, Grassin-Delyle S, Louedec L, Dupont S, Lamy E, Coggia M, Michel JB, Coscas R. An Experimental Study of Paclitaxel Embolisation During Drug Coated Balloon Angioplasty. Eur J Vasc Endovasc Surg. 2019 Apr;57(4):578-586. doi: 10.1016/j.ejvs.2018.11.019. Epub 2019 Mar 11. PMID 30871939
- [Background] Nakamura R, Torii S, Kato T, Kawasaki D. A Case of Vasculitis Due to Distal Particulate Embolization After Use of Drug-Coated Balloon. JACC Cardiovasc Interv. 2022 Jul 25;15(14):1486-1487. doi: 10.1016/j.jcin.2022.05.030. Epub 2022 Jun 29. No abstract available. PMID 35780056
- [Background] Torii S, Yahagi K, Mori H, Harari E, Romero ME, Kolodgie FD, Young B, Ragheb A, Virmani R, Finn AV. Biologic Drug Effect and Particulate Embolization of Drug-Eluting Stents versus Drug-Coated Balloons in Healthy Swine Femoropopliteal Arteries. J Vasc Interv Radiol. 2018 Jul;29(7):1041-1049.e3. doi: 10.1016/j.jvir.2018.02.006. Epub 2018 May 10. PMID 29754850
- [Background] Torii S, Jinnouchi H, Sakamoto A, Romero ME, Kolodgie FD, Virmani R, Finn AV. Comparison of Biologic Effect and Particulate Embolization after Femoral Artery Treatment with Three Drug-Coated Balloons in Healthy Swine Model. J Vasc Interv Radiol. 2019 Jan;30(1):103-109. doi: 10.1016/j.jvir.2018.07.025. Epub 2018 Dec 7. PMID 30527654
- [Background] Milewski K, Afari ME, Tellez A, Aboodi MS, Kim JS, Cheng Y, Conditt GB, McGregor JC, Yi GH, Stenoien M, Langanki D, Krueger CG, Kaluza GL, Granada JF. Evaluation of efficacy and dose response of different paclitaxel-coated balloon formulations in a novel swine model of iliofemoral in-stent restenosis. JACC Cardiovasc Interv. 2012 Oct;5(10):1081-8. doi: 10.1016/j.jcin.2012.06.012. PMID 23078739
- [Background] Vos NS, Fagel ND, Amoroso G, Herrman JR, Patterson MS, Piers LH, van der Schaaf RJ, Slagboom T, Vink MA. Paclitaxel-Coated Balloon Angioplasty Versus Drug-Eluting Stent in Acute Myocardial Infarction: The REVELATION Randomized Trial. JACC Cardiovasc Interv. 2019 Sep 9;12(17):1691-1699. doi: 10.1016/j.jcin.2019.04.016. Epub 2019 May 21. PMID 31126887
- [Background] Chen D, Yidilisi A, Zhang Y, Fang J, Zheng Y, Gao F, Li W, Zhou H, Chen Y, Lu D, Wang J, Jiang J. Fractional Flow Reserve-Guided Drug-Coated Balloon vs Drug-Eluting Stent for de Novo Non-Small Coronary Lesions. JACC Cardiovasc Interv. 2024 May 13;17(9):1182-1184. doi: 10.1016/j.jcin.2024.01.276. Epub 2024 Feb 21. No abstract available. PMID 38385923
- [Background] Shin ES, Ann SH, Balbir Singh G, Lim KH, Kleber FX, Koo BK. Fractional flow reserve-guided paclitaxel-coated balloon treatment for de novo coronary lesions. Catheter Cardiovasc Interv. 2016 Aug;88(2):193-200. doi: 10.1002/ccd.26257. Epub 2015 Oct 1. PMID 26423017
- [Background] Chung JH, Lee KE, Her AY, Lee JM, Doh JH, Nam CW, Koo BK, Shin ES. Comparison of fractional flow reserve and angiographic characteristics after balloon angioplasty in de novo coronary lesions. Int J Cardiovasc Imaging. 2019 Nov;35(11):1945-1954. doi: 10.1007/s10554-019-01649-y. Epub 2019 Jun 18. PMID 31214851
- [Background] Vrints C, Andreotti F, Koskinas KC, Rossello X, Adamo M, Ainslie J, Banning AP, Budaj A, Buechel RR, Chiariello GA, Chieffo A, Christodorescu RM, Deaton C, Doenst T, Jones HW, Kunadian V, Mehilli J, Milojevic M, Piek JJ, Pugliese F, Rubboli A, Semb AG, Senior R, Ten Berg JM, Van Belle E, Van Craenenbroeck EM, Vidal-Perez R, Winther S; ESC Scientific Document Group. 2024 ESC Guidelines for the management of chronic coronary syndromes. Eur Heart J. 2024 Sep 29;45(36):3415-3537. doi: 10.1093/eurheartj/ehae177. No abstract available. PMID 39210710
- [Background] Pijls NH, De Bruyne B, Peels K, Van Der Voort PH, Bonnier HJ, Bartunek J Koolen JJ, Koolen JJ. Measurement of fractional flow reserve to assess the functional severity of coronary-artery stenoses. N Engl J Med. 1996 Jun 27;334(26):1703-8. doi: 10.1056/NEJM199606273342604. PMID 8637515
- [Background] Ann SH, Balbir Singh G, Lim KH, Koo BK, Shin ES. Anatomical and Physiological Changes after Paclitaxel-Coated Balloon for Atherosclerotic De Novo Coronary Lesions: Serial IVUS-VH and FFR Study. PLoS One. 2016 Jan 29;11(1):e0147057. doi: 10.1371/journal.pone.0147057. eCollection 2016. PMID 26824602
- [Background] Guo S, Bi C, Wang X, Lv T, Zhang Z, Chen X, Yan J, Mao D, Huang W, Ye M, Liu Z, Xie X. Comparative efficacy of interventional therapies and devices for coronary in-stent restenosis: A systematic review and network meta-analysis of randomized controlled trials. Heliyon. 2024 Mar 8;10(6):e27521. doi: 10.1016/j.heliyon.2024.e27521. eCollection 2024 Mar 30. PMID 38496861
- [Background] Ahmad WAW, Nuruddin AA, Abdul Kader MASK, Ong TK, Liew HB, Ali RM, Mahmood Zuhdi AS, Ismail MD, Yusof AKM, Schwenke C, Kutschera M, Scheller B. Treatment of Coronary De Novo Lesions by a Sirolimus- or Paclitaxel-Coated Balloon. JACC Cardiovasc Interv. 2022 Apr 11;15(7):770-779. doi: 10.1016/j.jcin.2022.01.012. Epub 2022 Mar 16. PMID 35305906
- [Background] Ninomiya K, Serruys PW, Colombo A, Reimers B, Basavarajaiah S, Sharif F, Testa L, Di Mario C, Nerla R, Ding D, Huang J, Kotoku N, Kageyama S, Kageyama M, Sevestre E, Fezzi S, Dijkstra J, O'Leary N, Morel MA, Garg S, Cortese B, Onuma Y. A Prospective Randomized Trial Comparing Sirolimus-Coated Balloon With Paclitaxel-Coated Balloon in De Novo Small Vessels. JACC Cardiovasc Interv. 2023 Dec 11;16(23):2884-2896. doi: 10.1016/j.jcin.2023.09.026. Epub 2023 Oct 23. PMID 37877914
- [Background] Gitto M, Sticchi A, Chiarito M, Novelli L, Leone PP, Mincione G, Oliva A, Condello F, Rossi ML, Regazzoli D, Gasparini G, Cozzi O, Stefanini GG, Condorelli G, Reimers B, Mangieri A, Colombo A. Drug-Coated Balloon Angioplasty for De Novo Lesions on the Left Anterior Descending Artery. Circ Cardiovasc Interv. 2023 Dec;16(12):e013232. doi: 10.1161/CIRCINTERVENTIONS.123.013232. Epub 2023 Oct 24. PMID 37874646
- [Background] Jeger RV, Eccleshall S, Wan Ahmad WA, Ge J, Poerner TC, Shin ES, Alfonso F, Latib A, Ong PJ, Rissanen TT, Saucedo J, Scheller B, Kleber FX; International DCB Consensus Group. Drug-Coated Balloons for Coronary Artery Disease: Third Report of the International DCB Consensus Group. JACC Cardiovasc Interv. 2020 Jun 22;13(12):1391-1402. doi: 10.1016/j.jcin.2020.02.043. Epub 2020 May 27. PMID 32473887
- [Background] Unverdorben M, Kleber FX, Heuer H, Figulla HR, Vallbracht C, Leschke M, Cremers B, Hardt S, Buerke M, Ackermann H, Boxberger M, Degenhardt R, Scheller B. Treatment of small coronary arteries with a paclitaxel-coated balloon catheter in the PEPCAD I study: are lesions clinically stable from 12 to 36 months? EuroIntervention. 2013 Sep;9(5):620-8. doi: 10.4244/EIJV9I5A99. PMID 24058078
- [Background] Madhavan MV, Kirtane AJ, Redfors B, Genereux P, Ben-Yehuda O, Palmerini T, Benedetto U, Biondi-Zoccai G, Smits PC, von Birgelen C, Mehran R, McAndrew T, Serruys PW, Leon MB, Pocock SJ, Stone GW. Stent-Related Adverse Events >1 Year After Percutaneous Coronary Intervention. J Am Coll Cardiol. 2020 Feb 18;75(6):590-604. doi: 10.1016/j.jacc.2019.11.058. PMID 32057373
- [Background] Kufner S, Ernst M, Cassese S, Joner M, Mayer K, Colleran R, Koppara T, Xhepa E, Koch T, Wiebe J, Ibrahim T, Fusaro M, Laugwitz KL, Schunkert H, Kastrati A, Byrne RA; ISAR-TEST-5 Investigators. 10-Year Outcomes From a Randomized Trial of Polymer-Free Versus Durable Polymer Drug-Eluting Coronary Stents. J Am Coll Cardiol. 2020 Jul 14;76(2):146-158. doi: 10.1016/j.jacc.2020.05.026. PMID 32646563
- [Background] Capodanno D, Angiolillo DJ. Timing, Selection, Modulation, and Duration of P2Y12 Inhibitors for Patients With Acute Coronary Syndromes Undergoing PCI. JACC Cardiovasc Interv. 2023 Jan 9;16(1):1-18. doi: 10.1016/j.jcin.2022.10.023. PMID 36599574
- [Background] Neumann FJ, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO; ESC Scientific Document Group. 2018 ESC/EACTS Guidelines on myocardial revascularization. Eur Heart J. 2019 Jan 7;40(2):87-165. doi: 10.1093/eurheartj/ehy394. No abstract available. PMID 30165437
- [Background] Cortese B, Micheli A, Picchi A, Coppolaro A, Bandinelli L, Severi S, Limbruno U. Paclitaxel-coated balloon versus drug-eluting stent during PCI of small coronary vessels, a prospective randomised clinical trial. The PICCOLETO study. Heart. 2010 Aug;96(16):1291-6. doi: 10.1136/hrt.2010.195057. PMID 20659948
- [Background] Latib A, Colombo A, Castriota F, Micari A, Cremonesi A, De Felice F, Marchese A, Tespili M, Presbitero P, Sgueglia GA, Buffoli F, Tamburino C, Varbella F, Menozzi A. A randomized multicenter study comparing a paclitaxel drug-eluting balloon with a paclitaxel-eluting stent in small coronary vessels: the BELLO (Balloon Elution and Late Loss Optimization) study. J Am Coll Cardiol. 2012 Dec 18;60(24):2473-80. doi: 10.1016/j.jacc.2012.09.020. Epub 2012 Nov 14. PMID 23158530
- [Background] Jeger RV, Farah A, Ohlow MA, Mangner N, Mobius-Winkler S, Leibundgut G, Weilenmann D, Wohrle J, Richter S, Schreiber M, Mahfoud F, Linke A, Stephan FP, Mueller C, Rickenbacher P, Coslovsky M, Gilgen N, Osswald S, Kaiser C, Scheller B; BASKET-SMALL 2 Investigators. Drug-coated balloons for small coronary artery disease (BASKET-SMALL 2): an open-label randomised non-inferiority trial. Lancet. 2018 Sep 8;392(10150):849-856. doi: 10.1016/S0140-6736(18)31719-7. Epub 2018 Aug 28. PMID 30170854
- [Background] Tang Y, Qiao S, Su X, Chen Y, Jin Z, Chen H, Xu B, Kong X, Pang W, Liu Y, Yu Z, Li X, Li H, Zhao Y, Wang Y, Li W, Tian J, Guan C, Xu B, Gao R; RESTORE SVD China Investigators. Drug-Coated Balloon Versus Drug-Eluting Stent for Small-Vessel Disease: The RESTORE SVD China Randomized Trial. JACC Cardiovasc Interv. 2018 Dec 10;11(23):2381-2392. doi: 10.1016/j.jcin.2018.09.009. PMID 30522667
- [Background] Lassen JF, Burzotta F, Banning AP, Lefevre T, Darremont O, Hildick-Smith D, Chieffo A, Pan M, Holm NR, Louvard Y, Stankovic G. Percutaneous coronary intervention for the left main stem and other bifurcation lesions: 12th consensus document from the European Bifurcation Club. EuroIntervention. 2018 Jan 20;13(13):1540-1553. doi: 10.4244/EIJ-D-17-00622. PMID 29061550
- [Background] Latib A, Ruparelia N, Menozzi A, Castriota F, Micari A, Cremonesi A, De Felice F, Marchese A, Tespili M, Presbitero P, Sgueglia GA, Buffoli F, Tamburino C, Varbella F, Colombo A. 3-Year Follow-Up of the Balloon Elution and Late Loss Optimization Study (BELLO). JACC Cardiovasc Interv. 2015 Jul;8(8):1132-1134. doi: 10.1016/j.jcin.2015.04.008. No abstract available. PMID 26205451
- [Background] Cortese B, Bertoletti A. Paclitaxel coated balloons for coronary artery interventions: a comprehensive review of preclinical and clinical data. Int J Cardiol. 2012 Nov 1;161(1):4-12. doi: 10.1016/j.ijcard.2011.08.855. Epub 2011 Sep 28. PMID 21955612
- [Background] Wohrle J. Drug-coated balloons for coronary and peripheral interventional procedures. Curr Cardiol Rep. 2012 Oct;14(5):635-41. doi: 10.1007/s11886-012-0290-x. PMID 22825918
- [Background] Scheller B, Speck U, Abramjuk C, Bernhardt U, Bohm M, Nickenig G. Paclitaxel balloon coating, a novel method for prevention and therapy of restenosis. Circulation. 2004 Aug 17;110(7):810-4. doi: 10.1161/01.CIR.0000138929.71660.E0. Epub 2004 Aug 9. PMID 15302790
- [Background] Mehilli J, Dibra A, Kastrati A, Pache J, Dirschinger J, Schomig A; Intracoronary Drug-Eluting Stenting to Abrogate Restenosis in Small Arteries (ISAR-SMART 3) Study Investigators. Randomized trial of paclitaxel- and sirolimus-eluting stents in small coronary vessels. Eur Heart J. 2006 Feb;27(3):260-6. doi: 10.1093/eurheartj/ehi721. Epub 2006 Jan 9. PMID 16401670
- [Background] Togni M, Eber S, Widmer J, Billinger M, Wenaweser P, Cook S, Vogel R, Seiler C, Eberli FR, Maier W, Corti R, Roffi M, Luscher TF, Garachemani A, Hess OM, Wandel S, Meier B, Juni P, Windecker S. Impact of vessel size on outcome after implantation of sirolimus-eluting and paclitaxel-eluting stents: a subgroup analysis of the SIRTAX trial. J Am Coll Cardiol. 2007 Sep 18;50(12):1123-31. doi: 10.1016/j.jacc.2007.06.015. Epub 2007 Sep 4. PMID 17868802
- [Background] Park KH, Park SW, Hong MK, Kim YH, Lee BK, Park DW, Choi BR, Kim MJ, Park KM, Lee CW, Cheong SS, Kim JJ, Park SJ. Comparison of the effectiveness of sirolimus- and paclitaxel-eluting stents for small coronary artery lesions. Catheter Cardiovasc Interv. 2006 Apr;67(4):589-94. doi: 10.1002/ccd.20700. PMID 16547937
- [Background] Tanimoto S, Daemen J, Tsuchida K, Garcia-Garcia HM, de Jaegere P, van Domburg RT, Serruys PW. Two-year clinical outcome after coronary stenting of small vessels using 2.25-mm sirolimus- and paclitaxel-eluting stents: insight into the RESEARCH and T-SEARCH registries. Catheter Cardiovasc Interv. 2007 Jan;69(1):94-103. doi: 10.1002/ccd.20907. PMID 17139687
- [Background] Zhang X, Wang Q, Wang X, Xu X, Zhu J. [Comparison of limus-eluting stent with paclitaxel-eluting stent for patients with coronary small vessel disease:a systematic review and meta-analysis]. Zhejiang Da Xue Xue Bao Yi Xue Ban. 2017 May 25;46(3):305-314. doi: 10.3785/j.issn.1008-9292.2017.06.14. Chinese. PMID 29039175
- [Background] Katsanos K, Spiliopoulos S, Kitrou P, Krokidis M, Karnabatidis D. Risk of Death Following Application of Paclitaxel-Coated Balloons and Stents in the Femoropopliteal Artery of the Leg: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Am Heart Assoc. 2018 Dec 18;7(24):e011245. doi: 10.1161/JAHA.118.011245. PMID 30561254
- [Background] Bohme T, Noory E, Beschorner U, Macharzina R, Zeller T. The SELUTION SLR drug-eluting balloon system for the treatment of symptomatic femoropopliteal lesions. Future Cardiol. 2021 Mar;17(2):257-267. doi: 10.2217/fca-2020-0085. Epub 2020 Aug 20. PMID 32815739
- [Background] Costa RA, Mandal SC, Hazra PK, Chopda M, Chandra P, Damiani LP, Abizaid A, Hiremath S. Sirolimus-Coated Balloon With a Microsphere-Based Technology for the Treatment of De Novo or Restenotic Coronary Lesions. Cardiovasc Revasc Med. 2022 Dec;45:18-25. doi: 10.1016/j.carrev.2022.08.037. Epub 2022 Sep 5. PMID 36192319
- [Background] Madanchi M, Cioffi GM, Attinger-Toller A, Seiler T, Somm S, Koch T, Tersalvi G, Wolfrum M, Moccetti F, Toggweiler S, Kobza R, Levine MB, Garcia-Garcia HM, Bossard M, Cuculi F. Metal free percutaneous coronary interventions in all-comers: First experience with a novel sirolimus-coated balloon. Cardiol J. 2022;29(6):906-916. doi: 10.5603/CJ.a2022.0106. Epub 2022 Nov 17. PMID 36385601
- [Background] Spaulding C, Krackhardt F, Bogaerts K, Urban P, Meis S, Morice MC, Eccleshall S. Comparing a strategy of sirolimus-eluting balloon treatment to drug-eluting stent implantation in de novo coronary lesions in all-comers: Design and rationale of the SELUTION DeNovo Trial. Am Heart J. 2023 Apr;258:77-84. doi: 10.1016/j.ahj.2023.01.007. Epub 2023 Jan 13. PMID 36642225
- [Background] Rezkalla SH, Stankowski RV, Hanna J, Kloner RA. Management of No-Reflow Phenomenon in the Catheterization Laboratory. JACC Cardiovasc Interv. 2017 Feb 13;10(3):215-223. doi: 10.1016/j.jcin.2016.11.059. PMID 28183461
- [Background] Kloner RA, Dai W. Glycoprotein IIb/IIIa inhibitors and no-reflow. J Am Coll Cardiol. 2004 Jan 21;43(2):284-6. doi: 10.1016/j.jacc.2003.11.005. No abstract available. PMID 14736450
- [Background] Com-Nougue C, Rodary C, Patte C. How to establish equivalence when data are censored: a randomized trial of treatments for B non-Hodgkin lymphoma. Stat Med. 1993 Jul 30;12(14):1353-64. doi: 10.1002/sim.4780121407. PMID 8210831
- [Background] Hicks KA, Stockbridge NL, Targum SL, Temple RJ. Bleeding Academic Research Consortium consensus report: the Food and Drug Administration perspective. Circulation. 2011 Jun 14;123(23):2664-5. doi: 10.1161/CIRCULATIONAHA.111.032433. No abstract available. PMID 21670240
- [Background] Cutlip DE, Windecker S, Mehran R, Boam A, Cohen DJ, van Es GA, Steg PG, Morel MA, Mauri L, Vranckx P, McFadden E, Lansky A, Hamon M, Krucoff MW, Serruys PW; Academic Research Consortium. Clinical end points in coronary stent trials: a case for standardized definitions. Circulation. 2007 May 1;115(17):2344-51. doi: 10.1161/CIRCULATIONAHA.106.685313. PMID 17470709
- [Background] Thygesen K. 'Ten Commandments' for the Fourth Universal Definition of Myocardial Infarction 2018. Eur Heart J. 2019 Jan 14;40(3):226. doi: 10.1093/eurheartj/ehy856. No abstract available. PMID 30649367
- [Background] Moussa ID, Klein LW, Shah B, Mehran R, Mack MJ, Brilakis ES, Reilly JP, Zoghbi G, Holper E, Stone GW. Consideration of a new definition of clinically relevant myocardial infarction after coronary revascularization: an expert consensus document from the Society for Cardiovascular Angiography and Interventions (SCAI). J Am Coll Cardiol. 2013 Oct 22;62(17):1563-70. doi: 10.1016/j.jacc.2013.08.720. PMID 24135581
- [Background] Garcia-Garcia HM, McFadden EP, Farb A, Mehran R, Stone GW, Spertus J, Onuma Y, Morel MA, van Es GA, Zuckerman B, Fearon WF, Taggart D, Kappetein AP, Krucoff MW, Vranckx P, Windecker S, Cutlip D, Serruys PW; Academic Research Consortium. Standardized End Point Definitions for Coronary Intervention Trials: The Academic Research Consortium-2 Consensus Document. Circulation. 2018 Jun 12;137(24):2635-2650. doi: 10.1161/CIRCULATIONAHA.117.029289. PMID 29891620
- See also: SELUTION SLR™ 014 In-stent Restenosis — http://clinicaltrials.gov/study/NCT04280029
- See also: Non-Inferiority Clinical Trials — http://www.fda.gov/regulatory-information/search-fda-guidance-documents/non-inferiority-clinical-trials